CLINICAL TRIAL: NCT01285193
Title: A Randomized Controlled Trial to Treat Hypertension by Regularising and Slowing Breathing
Brief Title: Treating Hypertension With Breath Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Penang Hospital, Malaysia (Other Government)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Ng Kum Keong, Clinical Research Centre, Penang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT10-HPP-001; NMRR-10-686-6238 (Other: Ministry of Health Malaysia)
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Hypertension
Keywords: hypertension; high blood pressure; treatment; breath control; breathing exercise; audio CD
MeSH Terms: conditions — Hypertension | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breath control (Experimental): A music CD with sound cues is used to guide the subject to breathe in a regular and slower rate. This is practiced for at least 15 minutes a day over 2 months.
  Interventions: Behavioral: Breath control

INTERVENTIONS:
Behavioral: Breath control — A music CD with sound cues is used to guide the subject to breathe in a regular and slower rate. This is practiced for at least 15 minutes a day over 2 months.
  Other Names: breathing exercise; slow breathing

SUMMARY:
The purpose of this study is to determine if blood pressure can be reduced in hypertensive subjects by regularising and slowing their breathing. This may be a safe and affordable complementary treatment for hypertension.

DETAILED DESCRIPTION:
This is a randomised controlled trial in which hypertensive subjects allocated to receive either a CD with relaxation music or one with the same music plus certain sound cues to guide the listener on when to breathe. The subjects will continue with their normal medications and the intervention will last 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Patients with essential hypertension
* Systolic BP from 140 to 159 mm Hg
* Diastolic BP from 90 to 99 mm Hg
* On hypertensive medication for at least 3 months before the study
* Hypertensive medication unchanged during the 3 months before the study
* Patients able to fill in a log sheet

Exclusion Criteria:

* ischaemic heart disease
* congestive heart failure
* cardiac arrhythmias
* renal failure
* diabetes mellitus
* previous stroke
* major organ failure
* cigarette smoking
* respiratory diseases
* psychiatric disorders
* severe obesity (BMI >35 kg/m2)
* hearing impairment
* unable to operate a CD player or do not have access to a CD player
* arm circumference <22 cm. or >42 cm.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Diastolic blood pressure | 2 months
  Change in diastolic blood pressure from baseline to end value at 2 months.

SECONDARY OUTCOMES:
Systolic blood presure | 2 months
  Change in systolic blood pressure from baseline to end value at 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kum Keong Ng, MBBS, Principal Investigator — Clinical Research Centre, Penang Hospital
Locations (1):
- Ng Kum Keong, George Town, Pulau Pinang, Malaysia

REFERENCES:
- [Result] Grossman E, Grossman A, Schein MH, Zimlichman R, Gavish B. Breathing-control lowers blood pressure. J Hum Hypertens. 2001 Apr;15(4):263-9. doi: 10.1038/sj.jhh.1001147. PMID 11319675
- [Derived] Kow FP, Adlina B, Sivasangari S, Punithavathi N, Ng KK, Ang AH, Ong LM. The impact of music guided deep breathing exercise on blood pressure control - A participant blinded randomised controlled study. Med J Malaysia. 2018 Aug;73(4):233-238. PMID 30121686